CLINICAL TRIAL: NCT00125931
Title: Inpatient Clinical Trial Examining the Effects of Pentazocine on Manic Symptoms
Brief Title: Effects of Pentazocine on Manic Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Beth L. Murphy MD, PhD, Principal Investigator, Mclean Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005P-001260
Record Dates: First submitted 2005-08-01; First posted 2005-08-02 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; mania; manic state; opiate; kappa
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — talwin Nx; Pentazocine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pentazocine/Talwin (Experimental): Talwin NX
  Interventions: Drug: Talwin Nx

INTERVENTIONS:
Drug: Talwin Nx — Talwin NX 50mg po twice
  Other Names: Pentazocine

SUMMARY:
The opiate neurotransmitter system is thought to be involved in many abnormal mood states. Some researchers have suggested that changes in this system may trigger the switch to/from manic and depressive states in bipolar disorder. One problem with most of the currently available opiate medications is that they can produce addiction/dependence. A particular kind of opiate medication known as kappa-opiates may be able to produce changes in this system with much less risk of addiction. This study looks at Talwin (a combination of pentazocine and naloxone), a medication which affects the kappa and mu opiate systems. The study will examine whether two doses of Talwin affect manic symptoms in people who have been admitted to the hospital. This study will give more information about the involvement of the opiate system in bipolar disorder, and give important information for use in developing new treatments.

DETAILED DESCRIPTION:
Opiates have a long history of treating mood disorders. Some researchers have suggested that changes in this system may trigger the switch to/from manic and depressive states in bipolar disorder. The clinical use of opiate medications has been limited by their abuse/dependence potential. Studies of opiate receptor subtypes have raised the possibility that medications targeting the kappa/dynorphin system could be used to target mood symptoms with reduced/limited addiction potential. Rodent studies at Mclean indicate that kappa-agonists have pro-depressant effects and kappa-antagonists have anti-depressant effects. In addition, antimanic/antipsychotic medications regulate the activity of dynorphin cells. This study is a pilot open-label investigation using Talwin, a combination of pentazocine and naloxone. Pentazocine is a kappa agonist and mixed mu agonist. Two doses of Talwin will be given to acutely manic inpatients in a cumulative-dosing strategy. Measurements of manic symptoms will be conducted before, during, and after administration. This study will determine whether pentazocine has an immediate or sustained impact on acute mania symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Young Mania Rating Scale (YMRS) greater than 14
* Inpatient

Exclusion Criteria:

* History of opiate abuse/dependence
* Recent history of substance abuse
* Pregnancy
* Unstable medical issues
* Use of opiate medications for pain management

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth L Murphy, MD, PhD, Principal Investigator — Mclean Hospital

REFERENCES:
- [Background] Ma J, Ye N, Lange N, Cohen BM. Dynorphinergic GABA neurons are a target of both typical and atypical antipsychotic drugs in the nucleus accumbens shell, central amygdaloid nucleus and thalamic central medial nucleus. Neuroscience. 2003;121(4):991-8. doi: 10.1016/s0306-4522(03)00397-x. PMID 14580949
- [Background] Carlezon WA Jr, Beguin C, DiNieri JA, Baumann MH, Richards MR, Todtenkopf MS, Rothman RB, Ma Z, Lee DY, Cohen BM. Depressive-like effects of the kappa-opioid receptor agonist salvinorin A on behavior and neurochemistry in rats. J Pharmacol Exp Ther. 2006 Jan;316(1):440-7. doi: 10.1124/jpet.105.092304. Epub 2005 Oct 13. PMID 16223871
- [Background] Mague SD, Pliakas AM, Todtenkopf MS, Tomasiewicz HC, Zhang Y, Stevens WC Jr, Jones RM, Portoghese PS, Carlezon WA Jr. Antidepressant-like effects of kappa-opioid receptor antagonists in the forced swim test in rats. J Pharmacol Exp Ther. 2003 Apr;305(1):323-30. doi: 10.1124/jpet.102.046433. PMID 12649385
- [Background] Todtenkopf MS, Marcus JF, Portoghese PS, Carlezon WA Jr. Effects of kappa-opioid receptor ligands on intracranial self-stimulation in rats. Psychopharmacology (Berl). 2004 Apr;172(4):463-70. doi: 10.1007/s00213-003-1680-y. Epub 2004 Jan 16. PMID 14727002
- [Result] Cohen BM, Murphy B. The effects of pentazocine, a kappa agonist, in patients with mania. Int J Neuropsychopharmacol. 2008 Mar;11(2):243-7. doi: 10.1017/S1461145707008073. Epub 2007 Sep 26. PMID 17897484

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were 18-60 year old male and female individuals who were currently hospitalized.
Groups:
- Treatment Group: Open label group with pentazocine treatment.
Period: Overall Study
Arm/Group | Treatment Group
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Inpatients with manic symptoms.
Groups:
- Open Label: Open label treatment with pentazocine
Arm/Group | Open Label
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Mania Symptoms Using MACS
Description: Assessment of current mania symptoms using Mania Acute Change Scale (MACS). All 20 questions on the scale have a 0 (absent)-4(most severe) range for describing mania symptoms. The mean MACS score totals were reported, with the total ranging from 0-80. A higher total score indicates a greater number of symptoms and higher symptom intensity, while a smaller score indicates a lesser number of symptoms and higher lower intensity.
Time Frame: hourly for 6 hours after first dose of pentazocine; hour 0 is the baseline score and also when first dose of pentazocine was administered
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Open Label Group: Mania symptoms with pentazocine compared to baseline symptoms.
Arm/Group | Open Label Group
Number analyzed (Participants) | 10
units on a scale
  Hour 2 | 18.6 (8.9) [0 to 39]
  Hour 3 | 11.0 (6.9) [0 to 37]
Statistical Analysis 1: Comparison: Open Label Group; comparison of mean scores at hour 2 vs 3; Test type: Superiority or Other; p = 0.01, ANOVA

2. Secondary Outcome: YMRS Scores
Description: Assessment of current mania symptoms using YMRS. All questions have a 0 (absent)-4(most severe) range for describing mania symptoms. The mean YMRS scores were reported, with the total ranging from 0-44. A higher total score indicates a greater number of symptoms and higher symptom intensity, while a smaller score indicates a lesser number of symptoms and higher lower intensity.
Time Frame: Each morning of the three-day study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open Label Group
Number analyzed (Participants) | 10
units on a scale
  pre-treatment day | 23.6 (8.9)
  treatment day | 22.0 (6.9)
  post-treatment day | 12.7 (8.4)
Statistical Analysis 1: Comparison: Open Label Group; comparison of mean score on treatment vs post-treatment days; Test type: Superiority or Other; p = 0.01, t-test, 1 sided
Statistical Analysis 2: Comparison: Open Label Group; comparison of mean scores at pre-treatment vs treatment days; Test type: Superiority or Other; p = 0.4, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 3 days: pre-treatment day, treatment day, post-treatment day
Arm/Group | Open Label Group
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 9/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Group (N=10)
Sedation (Nervous system disorders) | 5 (5)
mild lightheadedness (Nervous system disorders) | 6 (6)
upset stomach (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of participants in open-label trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No